CLINICAL TRIAL: NCT00495248
Title: Well-being, Activity and Social Participation After Stroke/TIA. RCT-psycho Social Intervention Study.
Brief Title: Thriving, Activity and Social Participation After Stroke
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ullevaal University Hospital (Other)
Collaborators: The Royal Norwegian Ministry of Health (Other); The Norwegian Women´s Public Health Association (Other)
Responsible Party: Unni Sveen - PhD, Ullevaal University Hospital, Department of Geriatric Medicine
Organization: Oslo University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: UUS838
Record Dates: First submitted 2007-07-02; First posted 2007-07-03 (Estimated); Last update posted 2011-08-09 (Estimated); Status verified 2011-08

CONDITIONS: Stroke
Keywords: group intervention; stroke; senior centres; health promotion
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Behavioral: Group intervention inspired by Lifestyle Redesign
- 2 (Active Comparator)
  Interventions: Behavioral: Group intervention inspired by Lifestyle Redesign

INTERVENTIONS:
Behavioral: Group intervention inspired by Lifestyle Redesign — Group intervention inspired by Lifestyle Redesign
  Other Names: Lifestyle councelling
Behavioral: Group intervention inspired by Lifestyle redesign — Lifestyle programme once a week for two hours over an intervention period of 9 months
  Arms: 1

SUMMARY:
The aim of the study is to evaluate the effect of a group intervention programme for community dwelling elders with stroke or TIA.The intervention is inspired by a Lifestyle Redesign method developed in the USA. The study is conducted as a multi centre randomized controlled trial. Participants are recruited from five hospitals and the intervention is implemented at six to seven senior centres. The control group is offered physical activity at the senior centre once a week. The intervention group is offered the same with addition of the programme inspired by Lifestyle Redesign. The study will contribute to knowledge whether the intervention will promote social participation and thriving in daily life and prevent social isolation and depressive symptoms among community dwelling elders with stroke or TIA.

DETAILED DESCRIPTION:
Stroke is a common disease among older people. In Norway 60-70 000 people live with sequela after stroke. Depressive symptoms, anxiety and social isolation are occurring among 20 to 60 percent. Little is known about intervention for people with mild neurological symptoms who simultaneously perceive social isolation, depression and reduced satisfaction in their daily life after stroke. Lifestyle redesign (LR) is developed in the USA and is a health promoting group intervention programme with focus on the participants' exchange of experiences and involvement. The aim of the study is to evaluate the effect on thriving, activity and social participation of a group intervention program inspired by Lifestyle redesign for community dwelling persons with stroke. The study is conducted as a multicentre randomized controlled trial. Participants are recruited from five hospitals and the intervention is carried through at six to seven senior centres. The control group is offered a physical activity programme at the senior centre once a week. The intervention group is offered the same with the additional intervention programme also once a week. The study will contribute to knowledge whether this group intervention will promote social participation and thriving in daily life and prevent social isolation and depressive symptoms among community dwelling elders with stroke or TIA.

ELIGIBILITY:
Inclusion Criteria:

* oral and written consent
* age 65+
* clinical stroke ref WHO definition
* home-dwelling previous to stroke
* home-service less than twice a week previous to stroke
* Barthel ADL-index >14 of 20
* MMS >23 of 30
* be able to communicate evaluated by Ulleval aphasia screening test

Exclusion Criteria:

* reduced consent
* severe disease
* clinical contradictions evaluated by the responsible physician

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2007-01; Primary Completion 2009-09 (Actual); Study Completion 2011-09 (Estimated)

PRIMARY OUTCOMES:
SF-36 | Approximately 3 months after stroke-BASELINE, after 6 and 9 months

SECONDARY OUTCOMES:
Hospital Anxiety Depression Scale (HAD), Canadian Occupational Performance Measure (COPM), Trail making A and B, Timed up and go (TUG) | Approximately 3 months after stroke-BASELINE, after 6 and 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Unni Sveen, PhD, Study Director — Ullevaal University Hospital ,Medical division, research Unit 0407 Oslo Norway
Locations (1):
- Ullevaal University Hospital, Department of Geriatric Medicine, Research Unit, Oslo, Oslo County, Norway